CLINICAL TRIAL: NCT05570292
Title: Study of Effects of Preoperative Oral Domperidone on Gastric Residual Volume After Clear Fluid Ingestion in Patients Scheduled for Elective Surgeries: Prospective , Randomized ,Double Blinded Controlled Study
Brief Title: Study of Effects of Preoperative Oral Domperidone on Gastric Residual Volume After Clear Fluid Ingestion in Patients Scheduled for Elective Surgeries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU MS210/2022
Record Dates: First submitted 2022-10-02; First posted 2022-10-06 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Gastric Residual Volume
MeSH Terms: interventions — Domperidone; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Domperidone (Active Comparator)
  Interventions: Drug: Domperidone
- Folic acid (Placebo Comparator)
  Interventions: Drug: Folic acid

INTERVENTIONS:
Drug: Domperidone — ultrasound guieded assesment of gastric residual volume will be done 2 h after oral injestion of domperidone tablet
  Arms: Domperidone
Drug: Folic acid — ultrasound guieded assesment of gastric residual volume will be done 2 h after oral injestion of folic acid tablet
  Arms: Folic acid

SUMMARY:
General Anesthesia requires preoperative fasting according to specific instructions. Regarding Fasting Guidelines, The American Society of Anesthesiologists (ASA) recommends patients to fast from fatty food or meat eight hours prior to surgery, non-human milk or light meal for six hours prior, breast milk for four hours prior, and clear liquids including water, pulp-free juice, and tea without milk for two hours prior to the anesthetic. ASA fasting guidelines application represents the primary method to avoid aspiration as it ensures that stomach is empty before induction of anesthesia. These guidelines cannot be applied on all cases as in urgent or emergent situations or in morbidities associated with delayed gastric emptying, like Diabetes mellitus and some neurological disorders (

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* aged between 18-65 years
* who are categorized by ASA physical status as I or II
* undergoing elective surgeries under general anesthesia

Exclusion Criteria:

* Patients with known or suspected delayed gastric emptying (e.g. Diabetes mellitus) -psychiatric disorders
* hypersensitivity to the study medications
* peoples undergoing surgeries that associated with high incidence of Post operative nausea and vomiting (PONV) (e.g. Cholecystectomy, gynecological, ophthalmological, otorhinolaryngological, and laparoscopic surgeries).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
assess the effect of oral Domperidone preoperatively on gastric residual volume by ultrasound for patients undergoing elective surgeries under general anesthesia | first 2 hours preoperative
  patients will receive 400 ml of apple juice as a clear fluid, two hours preoperatively, and oral Domperidone tab or placebo tab

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt